CLINICAL TRIAL: NCT04201223
Title: The FLARE Skin Cancer Prevention Intervention for Children of Melanoma Survivors
Brief Title: Family Lifestyles, Actions, and Risk Education Intervention: Version 2
Acronym: FLARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Utah (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Yelena Wu, Assistant Professor, Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00114901; 133811-RSG-19-121-01-CPPB (Other Grant/Funding Number: American Cancer Society, Inc.)
Record Dates: First submitted 2019-11-26; First posted 2019-12-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Melanoma; Child
Keywords: Education; Prevention and Control; Behavioral Research
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLARE Intervention (Experimental): Participants will be randomized to receive an intervention that works with melanoma survivors and their children as a family unit to improve melanoma preventive behaviors.
  Interventions: Behavioral: FLARE Intervention
- Standard Education (No Intervention): Participants will be randomized to receive information on child sun protection that is publicly available.

INTERVENTIONS:
Behavioral: FLARE Intervention — [See arm/group descriptions]
  Arms: FLARE Intervention

SUMMARY:
The overall purpose of this study is to determine the efficacy of the Family Lifestyles, Actions, and Risk Education (FLARE) intervention in improving melanoma preventive behaviors. Parent-child dyads, consisting of survivors of melanoma and their children, will be randomly assigned to either receive the FLARE intervention or standard education. Once enrolled, each parent-child dyad will participate in this study for just over 1 year. Both conditions will receive three bi-weekly live intervention sessions (30 minutes per session) with an interventionist, and quarterly boosters via text or email.

DETAILED DESCRIPTION:
Enrollment

After parent-child dyads complete screening and informed consent/assent procedures, participants will be invited to complete an online baseline assessment. Following the baseline assessment, dyads will be randomized to receive either the FLARE intervention or standard education. After randomization, each dyad will receive a unique log-in to a secure study website that will be used to review didactic materials prior to each intervention session.

Intervention Sessions

Dyads will meet with an interventionist via remotely-delivered live session for their three intervention sessions. Intervention sessions will be scheduled every two weeks. After completion of the last remotely-delivered session, all parents will receive quarterly booster messages via text or email.

Study Assessments

Dyads will be asked to complete online assessments after consent is given (baseline) and within the 4 days prior to Session 3. A first post-intervention assessment will occur 4 weeks after the last intervention session is held. A second post-intervention assessment will occur 4 weeks later. The long-term follow-up assessment will take place 1-year post-baseline. Each assessment is expected to take 15-30 minutes. Parents will also receive a brief assessment via text or email (depending on parent preference) at monthly intervals between the second post-assessment and the 1-year post-baseline assessment, and in the summer months immediately following the 1-year post-baseline assessment. All assessments will be completed electronically.

ELIGIBILITY:
Inclusion Criteria:

Adults are eligible for this trial if they:

* Are at least 18 years old AND
* Have been diagnosed with melanoma at any time in their life AND
* Have at least one biological child between the ages of 8-17 years who is able to participate in the trial with them.

Children are eligible to participate with their parent if they:

* Are between the ages of 8-17 years AND
* Had at least 1 sunburn in the last 12 months AND
* Have at least one biological parent with a history of melanoma who can participate in the trial with them.

Exclusion Criteria:

Adults and children will be excluded from participation if they:

* Do not speak English OR
* Are unable to participate due to developmental delay OR
* Received testing for a mutation in CDKN2A/p16, including those who participated in a previous study where they received information on CDKN2A/p16.

Ages: 8 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Child Sunburn Occurrence Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), Monthly Assessment (Wk 18-41), 1-Year Follow-Up (Wk 52), Follow-Up 2 (Wk 56), Follow-Up 3 (Wk 60), Follow-Up 4 (Wk 64)
  We will examine whether sunburn occurrence decreased over time from pre- to post-intervention (Baseline through Post-Assessment 2), specifically whether the odds of sunburn occurrence are lower for FLARE compared to standard education. Additional analyses will compare sunburn occurrence between groups immediately post-intervention at Post-Assessment 1, and over the course of one year post-baseline. In all analyses, we will control for differences in sun exposure over time.
  "In the past (time period), how many times did you have a red OR painful sunburn that lasted a day or more?" Minimum value = 0; Maximum value = 5 or more; Lower scores indicate a better outcome.

SECONDARY OUTCOMES:
Skin Tone Assessed Via 11-Point Skin Color Palette | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/Standard deviation of the difference in skin tone between timepoints. Minimum value = 1; Maximum value = 11; Higher score indicates darker skin tone.
Sunscreen Application Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in sunscreen application occurrence between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you use a screen with an SPF of 30+?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Sunscreen Re-Application Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in sunscreen re-application occurrence between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you re-apply sunscreen after being outside for 2 hours, in the water, or sweating?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Long Sleeved Shirt Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in long sleeved shirt occurrence between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you wear a shirt with long sleeves?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Long Pants/Skirt Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in long pants/skirt occurrence between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you wear long pants or a long skirt?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Shade Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in shade occurrence between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you stay in the shade or under an umbrella?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Peak Hours Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in avoidance of peak hours between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you avoid being in the sun between 10:00AM-4:00PM?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Time Spent in the Sun to get Tan Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Session 3 (Wk 5-6), Post-Assessment 1 (Wk 8-11), Post-Assessment 2 (Wk 12-15), 1-Year Follow-Up (Wk 52)
  Mean/standard deviation of the difference in time spent in the sun to get tan between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you spend time in the sun in order to get a tan?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Wu, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Wu YP, Stump TK, Deboeck PR, Hay JL, Aspinwall LG, Boucher KM, Grossman D, Mooney K, Leachman SA, Smith KR, Brady HL, Hancock SE, Wankier AP, Tercyak KP. Sun protection, sunburn, tanning, and family factors among melanoma survivors and their minor children. J Health Psychol. 2025 Oct 9:13591053251378226. doi: 10.1177/13591053251378226. Online ahead of print. PMID 41067748

DOCUMENTS (1):
  • Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT04201223/ICF_001.pdf